CLINICAL TRIAL: NCT05603026
Title: Comparison of Hemodynamic Performance of Transcatheter Aortic Valve Replacement With Supra-Annular Self-Expanding Versus Balloon-Expandable Valves Assessed by Exercise Cardiovascular Magnetic Resonance
Brief Title: MRI in Transcatheter Aortic Valve Replacement Patients
Acronym: MRI-TAVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Guilherme Attizzani, MD, Physician, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20200834
Record Dates: First submitted 2022-10-24; First posted 2022-11-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVR; aortic stenosis; cardiac magnetic resonance; exercise cardiovascular magnetic resonance; magnetic resonance imaging; self-expanding valve; balloon-expandable valve; aortic bioprosthesis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TAVR using the self-expanding valve Evolut FX (Active Comparator): Transcatheter aortic valve replacement (TAVR) using the bioprosthesis Medtronic Evolut FX supra-annular self-expanding valve
  Interventions: Device: Self-expanding valve (Medtronic Evolut FX)
- TAVR using the balloon-expandable valve Sapien 3 Ultra RESILIA (Active Comparator): Transcatheter aortic valve replacement (TAVR) using the bioprosthesis Edwards Sapien 3 Ultra valve
  Interventions: Device: Balloon-expanding valve (Edwards Sapien 3 Ultra RESILIA)

INTERVENTIONS:
Device: Self-expanding valve (Medtronic Evolut FX) — Bioprothesis Medtronic Evolut FX supra-annular self-expanding valve
  Arms: TAVR using the self-expanding valve Evolut FX
Device: Balloon-expanding valve (Edwards Sapien 3 Ultra RESILIA) — Bioprosthesis Edwards Sapien 3 Ultra valve
  Arms: TAVR using the balloon-expandable valve Sapien 3 Ultra RESILIA

SUMMARY:
The hypothesis is that SEV result in superior valvular hemodynamics (more pronounced during exercise) and exercise capacity relative to BEV. Furthermore, the hypothesis is that stress CMR will be able to demonstrate differences in these hemodynamic parameters. CMR will also provide refined assessment of paravalvular leak and its impact on ventricular function and on clinical outcomes.

DETAILED DESCRIPTION:
Project Overview/Summary Transcatheter aortic valve replacement (TAVR) is an alternative to open heart surgery for the treatment of severe aortic stenosis, and has recently been approved for low surgical risk patients. This has resulted in a shifting of TAVR patient demographics to younger and more active individuals. It is, therefore, imperative to deliver excellent hemodynamics after valve replacement to enable patients to recover an active lifestyle with enhanced exercise capacity. Several studies, mostly conducted with resting echocardiogram have suggested self-expanding valves (SEV) Evolut R, Evolut PRO, Evolut PRO+ (Medtronic , Minneapolis, MN) are associated with favorable hemodynamics, which may allow for improved exercise capacity in active patients.

Currently, there are different TAVR valves are commercially available in the United States. The Sapien 3 valve (Edwards Lifesciences, Irvine, CA) is an annular, balloon expandable valve (BEV) and the Evolut PRO+ valve features a supra-annular design and is a SEV. A recent study utilizing resting echocardiogram demonstrated better hemodynamics of supra-annular SEV compared with BEV, mostly in patients with smaller annuli.

Cardiac magnetic resonance (CMR) has emerged as an important tool in the non-invasive assessment of patients with valvular heart disease. While CMR has been used for the diagnosis and quantification of valvular heart disease, there is a paucity of data on its use for the assessment of valvular hemodynamics in the post TAVR setting. Furthermore, it would be of utmost importance to understand how these devices perform during exertion. Of note, cardiac magnetic resonance techniques permit quantification of the myocardial extracellular volume fraction (ECV), representing a surrogate marker of reactive interstitial fibrosis, and late gadolinium enhancement (LGE), representing replacement fibrosis or scar. ECV and LGE have been independently linked with heart failure (HF) events.

Several studies have demonstrated that non-invasive CMR can be used to calculate non-invasive pressure-volume loops using cine imaging and non-invasive brachial blood pressure. This enables assessment of myocardial performance beyond LVEF. CMR-derived myocardial stroke work is a novel method allowing non-invasive assessment of total active myocardial performance, including both constructive and wasted myocardial work. Specifically, changes in LV stroke work have been shown to carry important prognostic information following TAVR.

Hypothesis The hypothesis is that SEV result in superior valvular hemodynamics (more pronounced during exercise) and exercise capacity relative to BEV. Furthermore, the hypothesis is that stress CMR will be able to demonstrate differences in these hemodynamic parameters. CMR will also provide refined assessment of paravalvular leak and its impact on ventricular function and on clinical outcomes.

STUDY DESIGN

Study Population There will be enrolled prospectively and retrospectively patients who have undergone TAVR at University Hospitals Cleveland Medical Center with different commercially available transcatheter valves and different sizes. It will then be screened all patients undergoing TAVR for a total of 90 patients.

All patients referred for TAVR will be considered for enrollment provided they meet the following inclusion and exclusion criteria. Inclusion criteria include all of the following: 1) Aortic valve stenosis with clinical indication for valve replacement decided by a dedicated heart team; 2) Planned transfemoral TAVR; 3) 18 years of age or older; 4) Able to give informed consent.

Exclusion criteria will include: 1) Patients with permanent pacemakers or implantable defibrillators; 2) Patients with non-MRI safe implants; 3) Severe claustrophobia; 4) Inability or contraindication to perform exercise bike stress test; 5) Arrhythmia which would prevent adequate cardiac gating, including atrial fibrillation; 6) Reduced left ventricular systolic function (<40%); 7) History of surgical aortic valve replacement or patients who undergo a valve-in-valve TAVR procedures; 8) Significant non-treated coronary artery disease.

Primary and Secondary Outcomes The co-primary endpoints will be analysed at 1-year follow up and will consist in: change in effective orifice area (EOA), mean gradient and peak gradient over time between valve types; and left ventricular stroke work.

Secondary outcomes will include: myocardial fibrosis; myocardial extra-cellular volume fraction; ability to perform stress CMR studies in post TAVR patient population, exercise capacity post TAVR, echocardiographic measures of valve and heart function, standard clinical outcomes of morbidity and mortality associated with TAVR.

Patient Enrollment, Treatment, and Follow-up Patients will be screened for inclusion/exclusion criteria as part of their pre-TAVR clinical evaluation. We will screen all patients undergoing TAVR for a total of 90 patients. There will be enrolled 45 patients to undergo TAVR and receive Sapien 3 BEV with two sizes (23 mm and 26 mm) and 45 patients to undergo TAVR with Evolut FX SEV in two available sizes (26 mm and 29 mm). All patients will be required to sign an informed consent. The choice for TAVR valve will be at the operator's discretion. Patients will be seen at 7- and 30-days post TAVR per routine clinical practice.

Baseline clinical parameters, procedural variables and the occurrence of MACE and bleeding events will be determined by history and corroborated by examining relevant medical records.

Transthoracic echocardiography will be performed immediately post TAVR, 1-day post TAVR and again at 30-days post TAVR as per standard clinical protocol. Patients will be treated with aspirin 81 mg daily and clopidogrel 75 mg daily for a minimum of 3 months, followed by aspirin 81 mg daily indefinitely thereafter.

MRI Imaging Protocol The first CMR will be performed up to three months prior to the TAVR procedure. Secondly, a stress CMR study will be performed 30-days (up to three months) post TAVR. Patients will have their EOA, valvular regurgitation, LV function, mean pressure gradient and peak pressure gradient assessed by standard MRI protocols. Patients will undergo an exercise stress MRI to assess exercise capacity, valve hemodynamics under stress and differences in hemodynamics between valve types. Finally, a follow up CMR will be performed 1-year after the TAVR, where it will be evaluated myocardial extracellular volume fraction and replacement fibrosis/scar in addition to the variables previously described.

CMR-Derived Non-invasive LV Pressure-Volume Loops It will be the able to calculate non-invasive pressure-volume loops using cine imaging and non-invasive brachial blood pressure. LVPV loops are derived non-invasively with ventricular-volume, heart rate and brachial pressure as inputs. LV stroke work is derived from the area of the generated pressure-volume loop.

MRI Stress Protocol The exercise MRI test will be performed on an MRI-compatible supine cycle ergometer that will be attached to the end of the MRI bed. Patients will be positioned on the gentry with a molding pad placed beneath them to help maintain patient position on the table during exercise for pre- and post-exercise scans. After initial imaging, the patient will remain supine on the table to complete the symptom-limited exercise stress test. Heart rate and blood pressure will be monitored continuously throughout exercise and during post-exercise scans. Immediately post-exercise, the patient will be placed back in the scanner for post-exercise.

Patient Safety Patients will be monitored for adverse events (AE) and serious adverse events (SAE). A data safety and monitoring board will be appointed to oversee and adjudicate these events. An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. Patients undergoing MRI and stress CMR will be screened for relevant contraindications by the research team at the time of their scan. SAE is an AE that results in death, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability, results in a congenital abnormality or birth defect, or is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above. The causality of SAEs (their relationship to all study treatments) will be assessed by the investigators. The following variables will be collected for each AE: 1) Type of AE, 2) Date and time when the AE started and stopped, 3) Whether the AE is serious or not, 4) Investigator causality rating against the investigational product, 5) Action taken with regard to investigational product, 6) Whether AE caused subject's withdrawal from the study, 7) Outcome. The following variables will be collected for each SAE: 1) Date AE met criteria for serious AE, 2) Date Investigator became aware of serious AE, 3) Reason AE is serious, 4) Date of hospitalization if applicable, 5) Date of discharge, if applicable, 6) Probable cause of death, if applicable, 7) Date of death, if applicable, 8) Autopsy performed, if applicable, 9) Causality assessment in relation to Study procedure(s), 10) Causality assessment in relation to other medication, 11) Description of AE.

Risks:

The only foreseeable risk of this study are:

1. Breach of confidentiality, which will be avoided by de-identifying patient data by name, and strictly guarding all data collected for the completion of the study.
2. Issues related to stress MRI: complications related to stress MRI, such as adverse reactions to drugs (ex. gadolinium), imaging features (ex. claustrophobia) or issues related to the stress induction (ex. fatigue, cardiac impairment) may occur, but will be explained prior to the image acquisition.

Benefits:

Through registry based analysis it will be isolated clinical determinants of morbidity and mortality, as well as the best clinical and procedural outcomes, which will inform best practices for TAVR procedures.

Statistical Analysis:

Continuous variables will be reported as median (interquartile range) and categorical variables as number (percentage). Cumulative survival free from outcomes will be assessed by Kaplan-Meier (KM) curves and Cox proportional hazard ratios will be calculated to create predictive and association models for the outcomes of interest. P-values of ≤0.05 will be considered statistically significant. Statistical analyses will be done using SAS, version 9.3 (SAS Institute, Cary, NC).

Data Safety Monitoring Plan:

The Principal Investigator will ensure that all the data is securely collected and stored in a password protected REDCap database. Each patient reviewed will be de-identified by a specific study number and names and MR numbers will not be used in the final statistical analysis. It will be ensured that after statistical analysis there is no means of connecting any patient reviewed to specific data associated with that patient.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve stenosis with clinical indication for valve replacement decided by a dedicated heart team;
* Planned transfemoral TAVR; 18 years of age or older;
* Able to give informed consent.

Exclusion Criteria:

* Patients with permanent pacemakers or implantable defibrillators;
* Patients with non-MRI safe implants;
* Severe claustrophobia;
* Inability or contraindication to perform exercise bike stress test;
* Arrhythmia which would prevent adequate cardiac gating, including atrial fibrillation;
* Reduced left ventricular systolic function (<40%);
* History of surgical aortic valve replacement or patients who undergo a valve-in-valve TAVR procedures;
* Significant non-treated coronary artery disease.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Effective orifice area (EOA) | Baseline, 30-days and 1-year
  Change in effective orifice area (EOA) assessed by CMR between baseline and 1-year follow up (cm2)
Mean gradient | 1-year
  Mean AV gradient assessed by CMR (mmHg)
Peak gradient | 1-year
  Mean AV gradient assessed by CMR (mmHg)

SECONDARY OUTCOMES:
Myocardial fibrosis | 1-year
  Myocardial fibrosis assessed by CMR (grams)
Myocardial extra-cellular volume fraction | 1-year
  Myocardial extra-cellular volume fraction assessed by CMR (Liters)
Stress CMR feasibility | 30-days
  Ability to perform stress CMR studies in post TAVR patient population (yes or no)
Exercise capacity post TAVR | 30-days
  Exercise capacity post TAVR assessed by CMR (METs)
Mean gradient by echo | 1-year
  Mean gradient assessed by transthoracic echocardiography (mmHg)
EOA by echo | 1-year
  Effective orifice area assessed by transthoracic echocardiography (cm2)
Ejection fraction by echo | 1-year
  Left ventricle ejection fraction assessed by transthoracic echocardiography (%)
Composite of morbidity and mortality associated with TAVR | 1-year
  Number of composite outcomes of morbidity and mortality associated with TAVR (number)

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Attizzani, MD, Principal Investigator — UH, Cleveland Medical Center; Sadeer Al-Kindi, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No